CLINICAL TRIAL: NCT00323284
Title: A Study of the Glaukos Trabecular Micro-Bypass Stent in Combination With Cataract Surgery in Open Angle Glaucoma Subjects.
Brief Title: A Study of the Trabecular Micro-bypass Stent in Combination With Cataract Surgery in Subjects With Open Angle Glaucoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Glaukos Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GC-003
Record Dates: First submitted 2006-05-06; First posted 2006-05-09 (Estimated); Results first posted 2012-10-04 (Estimated); Last update posted 2018-01-12 (Actual); Status verified 2016-03

CONDITIONS: Open-Angle Glaucoma
Keywords: Open angle; Glaucoma; Cataract; Surgery
MeSH Terms: conditions — Glaucoma, Open-Angle; Glaucoma; Cataract | interventions — Cataract Extraction; Phacoemulsification

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: IOP measurement
Oversight: Data Monitoring Committee: No

ARMS (2):
- A--iStent plus Cataract Surgery (Active Comparator): iStent plus Cataract Surgery
  Interventions: Device: iStent plus Cataract Surgery
- B--Cataract Surgery Only (Active Comparator): Cataract Surgery only
  Interventions: Procedure: Cataract surgery only

INTERVENTIONS:
Device: iStent plus Cataract Surgery — ab interno trabecular bypass stent surgery
  Other Names: iStent Surgery
  Arms: A--iStent plus Cataract Surgery
Procedure: Cataract surgery only — Cataract surgery only
  Other Names: Phacoemulsification
  Arms: B--Cataract Surgery Only

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of the iStent trabecular micro-bypass stent in reducing intraocular pressure (IOP) in subjects with open-angle glaucoma or ocular hypertension and co-existing cataract.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the safety and efficacy of the iStent trabecular micro-bypass stent in reducing intraocular pressure (IOP) in subjects with open-angle glaucoma or ocular hypertension and co-existing cataract. Pre-operative unmedicated baseline pressures will be compared with post operative values in both study arms.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with open-angle glaucoma (OAG) in the study eye. Pseudoexfoliative and pigmentary glaucoma are also acceptable diagnoses.
* Subject on at least one glaucoma medication
* Able and willing to attend follow up visits for two years post operative
* Able and willing to sign informed consent

Exclusion Criteria:

* Prior glaucoma procedures (eg trabeculectomy, viscocanalostomy, ALT, SLT, shunt implant, collagen implant, cyclo destructive procedures etc)
* Angle closure glaucoma
* Fellow eye already enrolled

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2005-06; Primary Completion 2009-07 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeff Wells, PharmD, MBA, Study Director — Glaukos Corporation
Locations (31):
- United States (31):
  - Assil Eye Institute, Beverly Hills, California
  - North Bay Eye Associates Inc, Petaluma, California
  - Ellison Ambulatory Care Center, Sacramento, California
  - Harvard Eye Associates, San Clemente, California
  - Shepard Eye Center, Santa Maria, California
  - Glaucoma Consultants of Colorado, Littleton, Colorado
  - Florida Eye Microsurgical Institute, Inc., Boynton Beach, Florida
  - The Center for Excellence in Eye Care, Miami, Florida
  - International Eye Center, Tampa, Florida
  - Clayton Eye Center, Morrow, Georgia
  - Indiana University, Indianapolis, Indiana
  - Stiles Eyecare Excellence, Overland Park, Kansas
  - The Eye Care Institute Building, Louisville, Kentucky
  - Williamson Nelson Eye Center, Baton Rouge, Louisiana
  - Kresge Eye Institute, Detroit, Michigan
  - Great Lakes Eye Care, Saint Joseph, Michigan
  - Chu Vision Institute, Edina, Minnesota
  - University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Discover Vision Centers, Independence, Missouri
  - Silverstein Eye Centers, Kansas City, Missouri
  - The Shepherd Eye Center, Las Vegas, Nevada
  - Glaucoma Consultants of Capital Region, Slingerlands, New York
  - Donald J. Digby and Associates, Greensboro, North Carolina
  - James Branch MD, Winston-Salem, North Carolina
  - Cinicinnati Eye Institute, Cincinnati, Ohio
  - Laurel Eye Center, Brookville, Pennsylvania
  - Wills Eye Hospital, Philadelphia, Pennsylvania
  - Associates in Ophthalmology, Pittsburgh, Pennsylvania
  - UPMC Eye Center, Pittsburgh, Pennsylvania
  - Southeast Texas Medical Association, L.L.P., Beaumont, Texas

REFERENCES:
- [Result] Samuelson TW, Katz LJ, Wells JM, Duh YJ, Giamporcaro JE; US iStent Study Group. Randomized evaluation of the trabecular micro-bypass stent with phacoemulsification in patients with glaucoma and cataract. Ophthalmology. 2011 Mar;118(3):459-67. doi: 10.1016/j.ophtha.2010.07.007. Epub 2010 Sep 15. PMID 20828829
- [Result] Craven ER, Katz LJ, Wells JM, Giamporcaro JE; iStent Study Group. Cataract surgery with trabecular micro-bypass stent implantation in patients with mild-to-moderate open-angle glaucoma and cataract: two-year follow-up. J Cataract Refract Surg. 2012 Aug;38(8):1339-45. doi: 10.1016/j.jcrs.2012.03.025. PMID 22814041

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study recruited subjects between April 2005 and February 2008. The main part of the study consisted of a randomized portion where subjects were randomized 1:1 to either iStent plus Cataract Surgery, or Cataract Surgery only. Following the randomized portion, addtional subjects were enrolled in a non-randomized portion.
Pre-assignment Details: Following screening, eligible subjects underwent a wash out of topical hypotensive medication prior to the baseline exam.
Period: 12 Months Follow-up
Arm/Group | A--iStent Plus Cataract Surgery | B--Cataract Surgery Only
Started | 116 | 123
Completed | 111 | 114
Not Completed | 5 | 9
Period: 24 Months Follow-up
Arm/Group | A--iStent Plus Cataract Surgery | B--Cataract Surgery Only
Started | 116 | 123
Completed | 98 | 101
Not Completed | 18 | 22

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | A--iStent Plus Cataract Surgery | B--Cataract Surgery Only | Total
Number analyzed (Participants) | 116 | 123 | 239
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 19 | 19 | 38
  >=65 years | 97 | 104 | 201
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.96 (7.66) | 72.88 (8.66) | 73.42 (8.11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 70 | 71 | 141
  Male | 46 | 52 | 98
Region of Enrollment [Number; unit: participants]
  United States | 116 | 123 | 239

OUTCOME MEASURES:

1. Primary Outcome: Intraocular Pressure (Measured in mm Hg) Less or Equal to 21 mm Hg on no Topical Hypotensive Meds
Description: Subjects with an intraocular pressure (IOP) less than or equal to 21 mm Hg without use of topical hypotensive medication at 12 months
Time Frame: 12 months
Population: Intent to treat analysis of all enrolled subjects using non-responder approach
Measure: Number (95% Confidence Interval); unit: percent of subjects achieving endpoint
Arm/Group | A--iStent Plus Cataract Surgery | B--Cataract Surgery Only
Number analyzed (Participants) | 116 | 123
percent of subjects achieving endpoint | 68 [60 to 77] | 50 [41 to 58]

2. Secondary Outcome: Efficacy
Description: Subjects with an intraocular pressure (IOP) reduction from baseline of greater than or equal to 20% without use of topical hypotensive medication at 12 months
Time Frame: 12 months
Population: Intent to treat population using non-responder approach
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | A--iStent Plus Cataract Surgery | B--Cataract Surgery Only
Number analyzed (Participants) | 116 | 123
percent | 64 [55 to 73] | 47 [38 to 56]

ADVERSE EVENTS:
Time Frame: Two years
Arm/Group | A--iStent Plus Cataract Surgery | B--Cataract Surgery Only
Serious Adverse Events (participants affected / at risk) | 1/116 | 1/123
Other Adverse Events (participants affected / at risk) | 27/116 | 42/123
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | A--iStent Plus Cataract Surgery (N=116) | B--Cataract Surgery Only (N=123)
Best Corrected Visual Acuity loss greater than 1 line at or after the 3 month visit (Eye disorders) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | A--iStent Plus Cataract Surgery (N=116) | B--Cataract Surgery Only (N=123)
Early post-op corneal edema (Eye disorders) | 9 (9) | 11 (11)
Posterior capsular opacification (Eye disorders) | 7 (7) | 12 (12)
Any BCVA loss greater than 1 line of vision at or after the 3 month visit (Eye disorders) | 7 (7) | 11 (11)
Blurry vision or visual disturbance (Eye disorders) | 4 (4) | 8 (8)

LIMITATIONS AND CAVEATS:
Open label given no way to mask treatment group to surgeon and visibility of iStent device upon gonioscopy.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days